CLINICAL TRIAL: NCT06036043
Title: Botulinum Toxin for Chronic Neuropathic Pain - an Interventional Open Label Study at the Interdisciplinary Pain Center, Zealand University Hospital
Brief Title: Botulinum Toxin for Chronic Neuropathic Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Region Zealand (Other)
Responsible Party: Principal Investigator, Rune Frederiksen, Principal Investigator, Region Zealand
Other Study IDs: RegionSealand
Record Dates: First submitted 2023-08-14; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Neuralgia; Chronic Pain
Keywords: Botulinum Toxin; chronic pain; neuropathic pain
MeSH Terms: conditions — Neuralgia; Chronic Pain | interventions — Botulinum Toxins, Type A; incobotulinumtoxinA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Intervention group: Patients treated with Botulinum Toxin
  Interventions: Drug: Botulinum toxin type A

INTERVENTIONS:
Drug: Botulinum toxin type A — The treatment will be administered either as a) subcutaneous infiltration with BoNT, covering the painful area, identified as allodynia during sensory examination, or b) perineural injection corresponding to the peripheral nerve(s) innervating the area where the pain is localized.
  1. 100 IU Xeomin is mixed with 4 ml NaCl. Injections are performed with a 1.5 cm spacing. Maximum of 40 injections (200 IU).
  2. 100 IU of botulinum toxin is mixed with 10 ml NaCl. For administration around multiple nerves, 50-100 IU per nerve (maximum 300 IU).
  The treatment will primarily be provided by the principal investigator, or an anesthesiologist specializing in nerve blocks.
  The specific method will be determined on an individual basis.
  If there is no effect after one to two treatments, the treatment will be considered ineffective and discontinued. A treatment interval of 3 months has been established in accordance with a previous larger study.
  Other Names: Xeomin

SUMMARY:
Treatment of peripheral neuropathic pain with Botulinum Toxin (BoNT) has showed promising results since the first study was released in 2001. Further research, however, is needed in order to strengthen the treatment, and a number of questions are unanswered. This includes which indication is the treatment the most effective, how should the treatment be administered, what is the duration of the effect? This study is a prospective interventional open label study, designed to assess the efficacy and safety of Botolinum toxin in the treatment of chronic neuropathic pain.

DETAILED DESCRIPTION:
Background:

There are eight randomized controlled trials investigating the effectiveness of BoNT for peripheral neuropathic pain. The indications in the studies include diabetic neuropathy, post-herpetic neuropathy, and peripheral nerve injury. Overall, the studies indicate a treatment effect that is significantly better than placebo. However, the studies are relatively small, their outcome measures vary, making comparison difficult, and there is considerable variation in the degree of pain reduction. The duration of the effect of BoNT treatment varies greatly and has not been systematically studied. The current evidence provides a promising background in the treatment of BoNT og neuropathic pain, but further research and documentation are needed.

At the Interdisciplinary Pain Center, Zealand University Hospital, BoNT treatment is already used for patients with neuropathic pain, who do not respond to 1. and 2. line treatments. This study will evaluate the efficacy of the treatment.

Method:

The objective of this study is to prospectively follow a one-year cohort and subsequently conduct a follow-up of 7 months (three treatments) for patients initiating BoNT treatment. The follow-up includes monitoring the treatment's effectiveness, duration, and recording adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* Condition of neuropathic pain verified by paraclinical examination or supported by underlying diseases (e.g., diabetes or herpes zoster).
* The condition is characterized by allodynia, hyperalgesia, and/or neuralgiform symptoms such as burning and stabbing pain.
* The affected area can be identified through objective examination with detection of disturbances in touch using cotton swabs, pin-prick, and/or vibration

Exclusion Criteria:

* Mixed etiology of pain not solely attributable to neuropathy (e.g., fibromyalgia and neuropathy or nociceptive pain and neuropathy).
* Contraindication to BoNT treatment (allergy to the toxin).
* Pregnancy.
* Diseases where BoNT treatment is contraindicated, such as motor neuron diseases and muscular dystrophy.
* Severe psychiatric disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic neuropathic pain
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximal pain intensity | At 28 days, 4 months, and 7 months after initiating treatment with BoNT type A (Xeomin®).
  Proportion of patients with clinically relevant reduction in maximum pain (last 24 hours) compared to baseline, assessed using the Numerical Rating Scale (NRS 0-10; Zero represents 'no pain at all' and the upper limit represents 'the worst pain ever possible'). A minimal important difference (MID) of NRS 1 is considered as clinically relevant.
pain intensity at rest | At 28 days, 4 months, and 7 months after initiating treatment with BoNT type A (Xeomin®)
  Proportion of patients with clinically relevant reduction in average pain at rest (last 24 hours) compared to baseline, assessed using the Numerical Rating Scale (NRS 0-10). A MID of NRS 1 is considered as clinically relevant.
Frequency of serious adverse events | Up to 7 months after initiating treatment
  Frequency of serious adverse events (according to ICH-GCP definition).
Frequency of serious adverse reactions | Up to 7 months after initiating treatment
  Frequency of serious adverse reactions (according to ICH-GCP definition).

SECONDARY OUTCOMES:
EuroQol-5 Dimension (EQ-5D) | At 28 days, 4 months, and 7 months after initiating treatment with BoNT type A (Xeomin®).
  Change in health-related quality of life (EQ-5D) compared to baseline. EQ-5D includes pain evaluation using the visual analogue scale (VAS 0-100; Zero represents 'no pain at all' and the upper limit represents 'the worst pain ever possible')
Neuropathic Pain Symptom Inventory (NPSI) | At 28 days, 4 months, and 7 months after initiating treatment with BoNT type A (Xeomin®).
  Change in neuropathic pain compared to baseline using the NPSI that evaluates 12 different symptoms according to a numerical rating scale from 0 to 10 (Zero represents 'no pain at all' and the upper limit represents 'the worst pain ever possible')
Onset and duration | At 28 days
  Time from treatment before onset of effect and duration of effect

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Peter Enggaard, MD, PHD, Study Director — Rigshospitalet, Denmark; Ole Mathiesen, MD, PHD, Study Director — University Hospital of Region Zealand
Locations (1):
- University Hospital of regions Zealand, Køge, Denmark

REFERENCES:
- [Background] Monheit GD, Pickett A. AbobotulinumtoxinA: A 25-Year History. Aesthet Surg J. 2017 May 1;37(suppl_1):S4-S11. doi: 10.1093/asj/sjw284. PMID 28388718
- [Background] Egeo G, Fofi L, Barbanti P. Botulinum Neurotoxin for the Treatment of Neuropathic Pain. Front Neurol. 2020 Aug 11;11:716. doi: 10.3389/fneur.2020.00716. eCollection 2020. PMID 32849195
- [Background] Datta Gupta A, Edwards S, Smith J, Snow J, Visvanathan R, Tucker G, Wilson D. A Systematic Review and Meta-Analysis of Efficacy of Botulinum Toxin A for Neuropathic Pain. Toxins (Basel). 2022 Jan 3;14(1):36. doi: 10.3390/toxins14010036. PMID 35051013
- [Background] Meyer-Friessem CH, Eitner LB, Kaisler M, Maier C, Vollert J, Westermann A, Zahn PK, Avila Gonzalez CA. Perineural injection of botulinum toxin-A in painful peripheral nerve injury - a case series: pain relief, safety, sensory profile and sample size recommendation. Curr Med Res Opin. 2019 Oct;35(10):1793-1803. doi: 10.1080/03007995.2019.1626228. Epub 2019 Jul 9. PMID 31148462
- [Background] Finnerup NB, Attal N, Haroutounian S, McNicol E, Baron R, Dworkin RH, Gilron I, Haanpaa M, Hansson P, Jensen TS, Kamerman PR, Lund K, Moore A, Raja SN, Rice AS, Rowbotham M, Sena E, Siddall P, Smith BH, Wallace M. Pharmacotherapy for neuropathic pain in adults: a systematic review and meta-analysis. Lancet Neurol. 2015 Feb;14(2):162-73. doi: 10.1016/S1474-4422(14)70251-0. Epub 2015 Jan 7. PMID 25575710
- [Background] Lippi L, de Sire A, Folli A, D'Abrosca F, Grana E, Baricich A, Carda S, Invernizzi M. Multidimensional Effectiveness of Botulinum Toxin in Neuropathic Pain: A Systematic Review of Randomized Clinical Trials. Toxins (Basel). 2022 Apr 27;14(5):308. doi: 10.3390/toxins14050308. PMID 35622555
- [Background] Attal N, de Andrade DC, Adam F, Ranoux D, Teixeira MJ, Galhardoni R, Raicher I, Uceyler N, Sommer C, Bouhassira D. Safety and efficacy of repeated injections of botulinum toxin A in peripheral neuropathic pain (BOTNEP): a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2016 May;15(6):555-65. doi: 10.1016/S1474-4422(16)00017-X. Epub 2016 Mar 2. PMID 26947719